CLINICAL TRIAL: NCT05733442
Title: Counseling for Harm Reduction and Retention in Medication-assisted Treatment - Cherokee Nation
Acronym: CHaRRM-CN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: University of Washington (Other); Cherokee Nation Health Services (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lonnie Nelson, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIRB 337; R33DA049376 (NIH)
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; harm reduction; medication assisted treatment; American Indian
MeSH Terms: conditions — Opioid-Related Disorders; Harm Reduction | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): The TAU condition will entail the current CNHS MAT program for OUD.
  Interventions: Other: Treatment as usual (TAU)
- CHaRRM-CN (Experimental): The CHaRRM-CN condition comprises changes and additions to TAU codesigned with a community advisory board and taking into account suggestions from MAT patients and community members impacted by OUD with the goal of improving MAT retention in culturally aligned and community-driven ways.
  Interventions: Other: CHaRRM-CN

INTERVENTIONS:
Other: Treatment as usual (TAU) — TAU entails medication to support patients' recovery (i.e., the partial opioid agonist, buprenorophine + naloxone/ Suboxone gel films), in-person case management and behavioral health intervention (i.e., in-person group and individual counseling), and referrals to other health care and behavioral health services.
  Arms: Treatment as Usual (TAU)
Other: CHaRRM-CN — The CHaRRM-CN intervention includes changes and additions to TAU to make MAT more culturally aligned (i.e., offering regular community-based, cultural programming; offering culturally aligned healing groups in the MAT program, such as Talking Circles and beading group) as well as lower barrier and incentivized (i.e., offering medication and behavioral health appointments via in-person, videoconference or telephone; offering harm-reduction groups in addition to abstinence-based groups; providing mailed and in-person pick-up options for buprenorphine prescriptions; conducting weekly chart reviews to ensure prescriptions and basic needs are continuously met; bimonthly, automated text outreach; contingency management supporting attendance at in-person or telehealth appointments).
  Arms: CHaRRM-CN

SUMMARY:
The goal of this randomized clinical trial is to test the efficacy of a program meant to enhance Counseling for Harm Reduction and Retention in MAT in Cherokee Nation (CHaRRM-CN). The main questions it aims to answer are whether CHaRRM-CN: improves retention of patients in MAT, decreases substance-related harm and illicit opioid use, and increases cultural connectedness.

After providing written, informed consent, participants will attend a baseline assessement and will then be randomized to either the CHaRRM-CN or treatment as usual group. For 6 months after randomization, participants will be exposed to CHaRRM-CN or treatment as usual. During that time, participants will also attend the 1-month, 3-month and 6-month follow-ups to track their progress through the programs.

After the 6 months of either treatment condition, investigators will compare the groups to see if they differ on retention, substance-use outcomes and Native enculturation.

DETAILED DESCRIPTION:
The opioid epidemic disproportionately impacts the American Indian (AI) population, which experiences an 88% higher prevalence of OUDs (1.5%) than the US general population (0.8%). The AI population is second only to non-Latinx whites in their experience of opioid overdose deaths (13.9 and 17.5 per 100,000, respectively). Fortunately, medication-assisted treatment (MAT; e.g., buprenorphine + naloxone) is highly effective for reducing opioid-related harm, including overdose, making it the gold-standard OUD treatment approach. A systematic review showed a median retention of 56% at the NIDA-recommended 12-month treatment length. However, most AI people with OUD do not attend traditional substance-use treatment (62%). This is concerning because treatment retention is strongly associated with a mortality rate reduction. Although no studies have documented OUD treatment outcomes specific to AI patients, research in Native communities has generally highlighted concerns about the cultural acceptability of the highly directive, Western medical substance-use treatment approaches (e.g., cognitive-behavioral therapy, 12-step programming) that are widely available. Further, previous research has indicated that AI patients with substance use disorders want greater representation of Native staff and better integration of culturally adapted approaches in the services they receive. Culturally adapted approaches to treatment are associated with reductions in use and associated harm. However, there are currently no evidence-based, culturally adapted counseling approaches for AI patients addressing MAT retention and opioid-related harm. Accordingly, the investigators are conducting a 2-phase R61/R33 development and evaluation project. The 2-year R61 Phase has been completed and entailed two parts. First, the investigators conducted a mixed methods inquiry to inform research methods and to create a community-specific, cultural adaptation of an existing, efficacious, harm-reduction counseling approach. Second, the investigators co-created and manualized the resulting Counseling for Harm Reduction and Retention in MAT at Cherokee Nation (CHaRRM-CN) together with a community advisory board comprising CNHS providers, staff, and patients as well as researchers from Cherokee Nation, Washington State University, and the University of Washington. The current, 3-year R33 Phase entails a 2-arm RCT (N=136) conducted within CNHS testing the efficacy of CHaRRM-CN in improving 6-month MAT retention, reducing substance-related harm and illicit opioid use, and increasing Native enculturation compared to a treatment-as-usual control condition.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Must be newly registered (within 4 weeks) in the CNHS MAT Program. (Prior patients can participate as long as their most recent treatment course was at least 6 months prior).
3. Must be willing to provide written informed consent to enroll in this study

Exclusion Criteria:

1. Refusal or inability to consent to participation in research. (The latter is assessed using the UCSD Brief Assessment of Capacity to Consent.)
2. Refusal or inability to consent and constituting a risk to the safety and security of other patients or staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
MAT retention | Month 6
  MAT program retention is defined by an active prescription for buprenorphine+naloxone with no gaps ≥ 30 days at month 6. This measure will dichotomously indicate whether participants have been retained in the MAT program (1) or not (0) at month 6.

SECONDARY OUTCOMES:
Substance-related harm | Baseline, month 1, month 3, month 6
  The Short Inventory of Problems will be used to collect data on substance-related harm in the past month. The range of possible scores on the single summary score is 0-45, and higher scores indicate a greater experience of substance-related harm. Change will be measured across the 4 points listed in the time frame.
Native enculturation | Baseline, month 1, month 3, month 6
  The Cultural Connectedness Scale - Short Version is a 10-item Likert type measure consisting of 3 dimensions: identity, traditions, and spirituality. Criterion validity was demonstrated with cultural connectedness dimensions adequately correlating with other indicators of wellness. Greater scores indicate greater cultural connectedness. Change will be measured across the 4 points listed in the time frame.
Native self-reliance | Baseline, month 1, month 3, month 6
  The Cherokee Self-Reliance Questionnaire includes 24, Likert-scale items that have been psychometrically validated in previous research.60,61 Consistent with the Cherokee self-reliance concept, the instrument comprises 3 factors: being responsible, disciplined, and confident. The higher the scale scores the higher the Native self-reliance. Change will be measured across the 4 points listed in the time frame.
Illicit Opioid Use | Baseline, month 1, month 3, month 6
  The Timeline Followback (TLFB) uses calendars for a retrospective evaluation of daily substance use. Meta-analyses have indicated the TLFB is a psychometrically sound way to detect substance use, including opioid use, across various populations and study designs. In the proposed study, the TLFB will be primarily used to assess use of illicit opioids. Change will be measured across the 4 points listed in the time frame.
ED visits | Baseline, month 6
  CNHS ED administrative data to assess number of visits to the ED both 6-months pre- and post-study enrollment. Change will be measured between the 2 points listed in the time frame.

OTHER OUTCOMES:
Health-related quality of life (HR-QoL) | Baseline, month 1, month 3, month 6
  The EuroQoL-5 Dimensional-5 Level (EQ-5D-5L) is a standardized 5-item, 5-point Likert-type measure of health-related QoL. This widely used, easily administered and psychometrically sound measure comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Additionally, a single, 100-point vertical visual analogue scale serves as a quantitative measure of participants' self-reported overall health status. The higher the scores, the higher the HR-QoL. This is an exploratory measure. Change will be measured across the 4 points listed in the time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie A Nelson, PhD, Principal Investigator — Washington State University; Susan E Collins, PhD, Principal Investigator — University of Washington; Ashley Lincoln, MSW, Principal Investigator — Cherokee Nation Health Services
Locations (2):
- United States (2):
  - Cherokee Nation Health Services, Tahlequah, Oklahoma
  - University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No